CLINICAL TRIAL: NCT05766670
Title: Intramedullary Calcium Sulfate Antibiotic Depot for Prevention of Open Fracture Related Infection: A Randomized Clinical Trial
Brief Title: Intramedullary Calcium Sulfate Antibiotic Depot
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: W81XWH-22-10937; W81XWH-22-10937 (Other: Department of Defense)
Record Dates: First submitted 2023-02-27; First posted 2023-03-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Open tíbia Fracture; Osteomyelitis Tibia; Tibial Fractures
Keywords: antibiotic depot
MeSH Terms: conditions — Tibial Fractures | interventions — Vancomycin; Gentamicins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intramedullary calcium sulfate antibiotic depot prior to Intramedullary nailing (IMN) placement (CS) (Other): The intramedullary calcium sulfate antibiotic depot will be mixed sterilely to include at minimum 20cc calcium sulfate powder mixed with 1g of vancomycin powder and 1.2g of tobramycin powder per 10cc of calcium sulfate.
  Interventions: Drug: Vancomycin Hydrochloride; Drug: Gentamicin
- Standard of care intramedullary nail (SN) (Other): Standard of care intramedullary nail
  Interventions: Other: Standard Intramedullary Nail

INTERVENTIONS:
Drug: Vancomycin Hydrochloride — The intramedullary calcium sulfate antibiotic depot will be mixed sterilely to include at minimum 20cc calcium sulfate powder mixed with 1g of vancomycin powder and 1.2g of tobramycin powder per 10cc of calcium sulfate.
  Other Names: antibacterial prescription medicine
  Arms: Intramedullary calcium sulfate antibiotic depot prior to Intramedullary nailing (IMN) placement (CS)
Drug: Gentamicin — The intramedullary calcium sulfate antibiotic depot will be mixed sterilely to include at minimum 20cc calcium sulfate powder mixed with 1g of vancomycin powder and 1.2g of tobramycin powder per 10cc of calcium sulfate.
  Other Names: injection is used to treat certain serious infections that are caused by bacteria such as meningitis
  Arms: Intramedullary calcium sulfate antibiotic depot prior to Intramedullary nailing (IMN) placement (CS)
Other: Standard Intramedullary Nail — Standard Intramedullary Nail
  Other Names: metal rod that is inserted into the medullary cavity of a bone and across the fracture in order to provide a solid support for the fractured bone
  Arms: Standard of care intramedullary nail (SN)

SUMMARY:
The goal of this randomized clinical trial is to study the best treatment for open lower leg fractures to prevent infection. The main questions it aims to answer is if treating tibia fracture patients with a calcium sulfate antibiotic depot is better at preventing infection that the standard of care.

DETAILED DESCRIPTION:
This research is a randomized clinical trial aimed to reduce the frequency of fracture related infections following open tibia fracture. The proposed test methods for infection reduction is use of an antibiotic depot placed inside the bone at the time of final fracture treatment. This is in addition to standard of care wound care, fracture fixation with intramedullary nailing, and peri-operative systemic antibiotics.

This prospective randomized clinical trial will compare outcomes between patients treated with an antibiotic depot placed inside the bone at the time of final fracture fixation and those treated with traditional standard of care intramedullary nailing.

The target population for the proposed study is patients with severe open tibia fractures (Type II or III) who require definitive fixation with intramedullary nail recruited form one of the participating sites during the index hospitalization.

One group will be treated prophylactically suing a calcium sulfate antibiotic depot at the time of definitive fixation, while the second group will be treated with a standard of care intramedullary nail without the antibiotic depot.

Participants will be followed for 12 months (data capture includes patient interviews and clinical data capture from the treatment team and medical record at baseline, 6 weeks, 3 months, 6 months, and 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Type II or III open tibia fracture requiring definitive fixation with intramedullary nail

Exclusion Criteria:

* Less than 18 years of age
* Allergy to vancomycin or tobramycin
* Hypercalcemia
* Unable to speak English or Spanish
* No email, phone, or other point of contact
* Pregnant and lactating women
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 497 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who develop deep surgical site infection (SSI) | Month 12
  Number of participants in each group who develop surgical site infection (SSI) as defined by the criteria establish by the Centers for Disease Control and Prevention (CDC). The CDC criteria define deep as occurring within 30 or 90 days after the procedure. However, we will continue to follow patients for 12 months and document any infections and other complications during this period.

SECONDARY OUTCOMES:
Number of Participants who Return to the Operating Room (OR) | Month 12
  Number of Participants who Return to the Operating Room (OR)
Percentage of Union | week 6, month 3, month 6 and month 12
  Union is the gradual process of bone regeneration after a fracture. Percentage of Union, as determined by the treating surgeon, will be assessed via radiographs. Recorded by surgeon as yes/no answers.
Time to Union | week 6, month 3, month 6 and month 12
  Captured in days
Radiographic Union Scale in Tibial fractures (RUST) score | week 6, month 3, month 6, and month 12
  The RUST score ranges from a minimum score of 4 (definitely not healed) to a maximum score of 12 (completely healed). The final x-ray obtained within a 12-month period following injury will be uploaded to REDCap for review by a blinded panel of investigators from participating sites.
Presence of drainage from incision and wounds | week 6, month 3, month 6 and month 12
  When present, patients will be asked to document the duration of drainage. Duration will be treated as a continuous variable with 7 days of drainage categorized as "persistent drainage".
Average Time to Return to Work/Duty | week 6, month 3, month 6 and month 12
  number of days
International Physical Activity Questionnaire (IPAQ) | Baseline, 3 month, 6 month, 12 month
  IPAQ measures the total amount of physical activity completed in a 7 day period by calculating the minutes per week in in each physical activity level domain (walking, moderate and vigorous) by a metabolic equivalent energy (MET) expenditure estimate.
  Walking = 3.3 x number of walking minutes x number of walking days Moderate activity= 4.0 x number activity minutes x number of days Vigorous activity = 8 x number of activity minutes x number of days Total = Walking MET-min/wk+moderate MET-min/wk+vigorous MET-min/wk
PROMIS-29 Subscale--Physical Function | week 6, month 3, month 6 and month12
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. The sum of the PROMIS results in the raw score, which lies between 4 and 20 - Higher scores means higher physical function; lower scores represent lower physical function
PROMIS-29 Subscale--Physical Function: Anxiety | week 6, month 3, month 6 and month12
  The PROMIS-29 scales will be scored using a T-score metric method. The PROMIS Anxiety item banks assess self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of anxiety; lower scores represent lower level of anxiety
PROMIS-29 Subscale--Depression | week 6, month 3, month 6 and month12
  The PROMIS-29 scales will be scored using a T-score metric method. For each scale, respondents are asked how often in the past 7 days they have experienced specific depression symptoms, using a 5-point ordinal rating scale of "Never," "Rarely," "Sometimes," "Often," and "Always." A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of depression; lower scores represent lower level of depression
PROMIS-29 Subscale--Fatigue | week 6, month 3, month 6 and month12
  The PROMIS-29 scales will be scored using a T-score metric method. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like fatigue, a T-score of 60 is one SD worse than average. By comparison, a fatigue T-score of 40 is one Standard Deviation better than average. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of fatigue. Mean fatigue scores in the four study samples ranged from 18.5 to 22.8 on the PROMIS (PROMIS) Fatigue-Short Form (F-SF) (potential range 7-35); from 14.8 to 47.8 on the MFSI-SF (potential range 24-86); and from 3.6 to 6.6 on the BFI (potential range 0-10).
PROMIS-29 Subscale--Sleep Disturbance | week 6, month 3, month 6 and month12
  The PROMIS-29 scales will be scored using a T-score metric method. The PROMIS Sleep Disturbance instruments assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of sleep disturbance. Total score is the sum of the seven subscale scores (ie, quality of sleep, quantity of sleep, sleep onset latency, midsleep awakenings, early awakenings, medications for sleep, excessive daytime sleepiness) that can range from 0 (no disturbance) to 147 (extreme sleep disturbance).
PROMIS-29 Subscale--Pain Interference | week 6, month 3, month 6 and month12
  The PROMIS-29 scales will be scored using a T-score metric method. PROMIS Pain Intensity T-scores from 20-55 are considered within normal limits, 55-60 is mild, 60-70 is moderate, and 70+ is severe. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of pain interference. PROMIS Pain Interference (PROMIS-PI) scale measures the extent to which pain hinders an individual's engagement with physical, mental, cognitive, emotional, recreational, and social activities.
PROMIS-29 Subscale--Ability to Participate in Social Roles and Activities | week 6, month 3, month 6 and month12
  The PROMIS-29 scales will be scored using a T-score metric method. Social function is defined by PROMIS as involvement in, and satisfaction with, one's usual social roles in life's situations and activities. These roles may exist in marital relationships, parental responsibilities, work responsibilities and social activities. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher ability to participate in social roles and activities.
Veterans RAND 12 Item Health Survey (VR-12) Domain --General Health | week 6, month 3, month 6 and month12
  The VR-12 is a measure of global health that correspond to seven domains. Together, these items are summarized into a Physical Component Score and a Mental Component Score. The VR-12 is a patient-reported instrument from which physical and mental health component summary scores (PCS and MCS) are derived. The PCS and MCS are normalized using TScore and are on a 0-100 scale. The interpretation is based on a population mean of 50 and standard deviation of 10. Higher scores represent a better outcome. The VR-12 items assess physical functioning, role limitations due to physical or mental health problems, pain, energy, mental health, social functioning, and general health.
Veterans RAND 12 Item Health Survey (VR-12) Domain--Physical Functioning | week 6, month 3, month 6 and month12
  The VR-12 is a measure of global health that correspond to seven domains. Together, these items are summarized into a Physical Component Score and a Mental Component Score. The VR-12 is a patient-reported instrument from which physical and mental health component summary scores (PCS and MCS) are derived. The PCS and MCS are normalized using TScore and are on a 0-100 scale. The interpretation is based on a population mean of 50 and standard deviation of 10. Higher scores represent a better outcome. The VR-12 items assess physical functioning, role limitations due to physical or mental health problems, pain, energy, mental health, social functioning, and general health.
Veterans RAND 12 Item Health Survey (VR-12) Domain--Role Limitations | week 6, month 3, month 6 and month12
  The VR-12 is a measure of global health that correspond to seven domains. Together, these items are summarized into a Physical Component Score and a Mental Component Score. The PCS and MCS are normalized using TScore and are on a 0-100 scale. The interpretation is based on a population mean of 50 and standard deviation of 10. Higher scores represent a better outcome.
Veterans RAND 12 Item Health Survey (VR-12) Domain--Pain | week 6, month 3, month 6 and month12
  The VR-12 is a measure of global health that correspond to seven domains. Together, these items are summarized into a Physical Component Score and a Mental Component Score. The PCS and MCS are normalized using TScore and are on a 0-100 scale. The interpretation is based on a population mean of 50 and standard deviation of 10. Higher scores represent a better outcome.
Veterans RAND 12 Item Health Survey (VR-12) Domain--Fatigue | week 6, month 3, month 6 and month12
  The VR-12 is a measure of global health that correspond to seven domains. Together, these items are summarized into a Physical Component Score and a Mental Component Score. The PCS and MCS are normalized using TScore and are on a 0-100 scale. The interpretation is based on a population mean of 50 and standard deviation of 10. Higher scores represent a better outcome.
Veterans Rand 12 Item Health Survey (VR-12) Domain --Social Functioning | week 6, month 3, month 6 and month12
  The VR-12 is a measure of global health that correspond to seven domains. Together, these items are summarized into a Physical Component Score and a Mental Component Score. The PCS and MCS are normalized using TScore and are on a 0-100 scale. The interpretation is based on a population mean of 50 and standard deviation of 10. Higher scores represent a better outcome.
Veterans Rand 12 Item Health Survey (VR-12) Domain--Mental Health | week 6, month 3, month 6 and month12
  The VR-12 is a measure of global health that correspond to seven domains. Together, these items are summarized into a Physical Component Score and a Mental Component Score. The PCS and MCS are normalized using TScore and are on a 0-100 scale. The interpretation is based on a population mean of 50 and standard deviation of 10. Higher scores represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel B Seymour, PhD, Principal Investigator — Wake Forest University Health Sciences; Jessica Rivera, MD, Principal Investigator — Louisiana State University Health Science Center
Locations (10):
- United States (10):
  - Cedars-Sinai, Los Angeles, California
  - Atrium Health Navicent The Medical Center, Macon, Georgia
  - University of Kentucky, Lexington, Kentucky
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Atrium Health Carolinas Medical Center, Charlotte, North Carolina
  - Atrium Health Cabarrus, Concord, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Pennsylvania State University, Hershey, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Valley Health, Winchester, Virginia

IPD SHARING:
Plan to Share IPD: No